CLINICAL TRIAL: NCT01490606
Title: A Comparative, Non Randomized Trial of Knee Osteoarthritis (OA) Project Treatment Versus Conventional Physical Therapy in the Treatment of Knee OA Patients
Brief Title: Knee Osteoarthritis (OA) Project Treatment Versus Conventional Physical Therapy in the Treatment of Knee OA Patients
Acronym: OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Shemtov Fatal, physical therapist, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC11191/2011KCTIL
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- knee OA project (Experimental): 12 sessions of PT, 6 INDIVIDUAL AND 6 GROUP TREATMENTS
  Interventions: Other: knee OA project; Other: conventional PT
- conventional PT (No Intervention)

INTERVENTIONS:
Other: knee OA project — physical therapy in "OA Knee project", total of 12 sessions, 6 group therapies amd 6 one on one therapy.
  Arms: knee OA project
Other: conventional PT — 12 SESSIONS OF CONVENTIONAL PHYSICAL THERAPY
  Arms: knee OA project

SUMMARY:
A. Background.

Patients with osteoarthritis (OA) of the knee, suffer from a combination of pain, stiffness, joint instability, swelling and muscles weakness. This leads to decrease in quality of life, Active Daily living (ADL) and increase of medical services consumption in the community. OA of the knee, Is one of the world's common musculoskeletal disorder (18% among women and 10% among men). 80% of patients with OA of the knee suffer from decrease in mobility and 20% of them suffer an inability to perform everyday activities.

Physical therapy training includes exercises for OA patients (Mild to Severe degree) is the cornerstone of non medicinal treatment. This training aimed to pain reduction, improved functioning and participation in family and working social life. Physical training with exercises can enhance physical capabilities such as: muscular strength, range of motion, balance, proprioception and cardiovascular performance. Other benefits are improving mobility, reducing risk of falls and body weight and improvement in psychological condition.

B. Purpose

The purpose of this research is to check the effectiveness of treatment in the framework of "knee Osteoarthritis project" compared to conventional Physical therapy in physical functioning, pain and quality of life scales, among patients over the age of 60 who suffer from OA of the knee .

C. Research method

A comparative non blinded, clinical trial will be conducted. This research will include 60 independent patients divided into equal groups: Intervention group will be trained in "knee Osteoarthritis project" (in which patients receive 6 individual treatments and 6 Group treatments). Control group will be treated with conventional physical therapy, which includes 12 individual treatments. Effect of the treatment will be evaluated by: 1. WOMAC questionnaire- used to evaluate function and pain. 2. EQ-5D questionnaire for evaluating the quality of life. 3. Time up and go test- a Common functional test. This Questionnaires and test will be Performed before and after the study.

D. Study hypothesis

Physical therapy treatment within the framework of "knee Osteoarthritis project" is favor than the treatment of the conventional Physical therapy. Therefore the investigators expect much improvement in terms of pain, physical functioning and quality of life among intervention group compared to control groups.

DETAILED DESCRIPTION:
This research is divided into o Intervention and control groups. Research Population is 60 Patients (30 patients to each arm), aged 60 and above suffering from OA of the knees and admitted to physical therapy .Intervention group patients were treated by the concept of "Knee Osteoarthritis Project". This was first applied in middle of 2010 and its effectiveness was never tested.

The main idea was to make patients more active, to encourage them to do exercise at home, increase their motivation and self efficacy. In addition, patients received prescription for TENS device (Transcutaneous electrical nerve stimulator) for home use.

Individual sessions include: muscle strengthening, proprioception exercise, taping, soft tissue stretching, joint and soft tissue mobilization, electrotherapy, aerobic exercise (bicycle, treadmill), functional exercise. Group session include: muscle strengthening, stairs exercise, balance exercise and education about the disease and treatment (lecture about knee OA and recommendations for changes in life style).

In Intervention group were given 12 session. 6 individual treatments and 6 group treatments Control group patients were given 12 individual sessions of conventional physical therapy.

The Outcome measures that were mention above will be performed in the beginning and the end of 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

* 60+ years old independent men and women,who suffer from OA in the knee and was referred to Physiotherapy.
* ability to write and read properly in Hebrew

Exclusion Criteria:

* OA secondary to systematic disease (Rheumatoid arthritis)
* steroids injections to the knee in the past 3 months.
* orthopaedic surgery to lower limbs.
* neurological deficit.
* symptomatic OA in the hip or ankle

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Time up and go test | On the first week- first session of PT and on last session- 12 weeks Average
  Patient sits on a chair with handles. by order "go", patient will stand up and walk 3 meters forward circle a Conus and return to the chair. a time watch will count time.
WOMAC questionaire | On the first week- first session of PT and on last session- 12 weeks Average
EQ-5D questionaire | On the first week- first session of PT and on last session- 12 weeks Average

SECONDARY OUTCOMES:
Body Mass index | Up to the first week- on the first session of PT

CONTACTS AND LOCATIONS:
Overall Officials: Yair Barzilai, M.D., Principal Investigator — Clalit health service, Israel
Locations (1):
- Clalit Health Service, Jerusalem, Israel, Israel